CLINICAL TRIAL: NCT04494672
Title: Improving Intramedullary Nailing of Proximal Femoral Fractures Through a Navigation Assisted Technique: a Double Blinded Randomized Control Trial
Brief Title: A Study to Verify if the Surgery for the Proximal Femur Fracture Can be Improved With the Help of a Navigation System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Candrian (Other)
Responsible Party: Sponsor-Investigator, Christian Candrian, Prof. Dr. Med., Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORL-ORT-015
Record Dates: First submitted 2020-07-21; First posted 2020-07-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Femoral Fracture
MeSH Terms: conditions — Femoral Fractures | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intramedullary nailing with ADAPT system (arm-A) (Experimental): A commercial product, namely ADAPT will be used as investigation product in arm-A
  Interventions: Procedure: Intramedullary nailing with ADAPT system
- Intramedullary nailing without ADAPT system (arm-B) (Active Comparator): No aid in performing intramedullary nailing for proximal femoral fractures will be implemented in arm-B
  Interventions: Procedure: Intramedullary nailing without ADAPT system

INTERVENTIONS:
Procedure: Intramedullary nailing with ADAPT system — Stryker ADAPT®system (ADAPT, Stryker Leibinger GmbH & Co. KG, Freiburg, Germany) is a computer navigation system which can reconstruct a 3D model of the femoral head from the positional information oriented by bidirectional fluoroscopic views. ADAPT shows the distance from the tip of the screw to the surface of the femoral head, tip-to-head-surface distance (TSD), and tip-apex distance (TAD) intraoperatively
  Arms: Intramedullary nailing with ADAPT system (arm-A)
Procedure: Intramedullary nailing without ADAPT system — Intramedullary nailing without ADAPT system
  Arms: Intramedullary nailing without ADAPT system (arm-B)

SUMMARY:
The ADAPT system is a software that calculate a virtual 3D reconstruction of the femoral head without additional radiation. It automatically detects the used implant and its position relative to the femoral head, helping the surgeon to achieve an optimal proximal screw positioning in the femoral head. The investigators want to verify if with the addition of the ADAPT system the investigators can improve screw placement and reduce surgery time and radiation exposure.

DETAILED DESCRIPTION:
This study is a 2-arm randomized controlled trial comparing intramedullary nailing of proximal fracture of the femur (AO classified as 31 A1.3 , 31 A2.1, 31 A2.2 31 A2.3, 31 A3.1, 31 A3.2, 31 A3.3) performed with the ADAPT system (arm-A) and those performed without (arm-B).

The ADAPT system has been developed with the aim to reduce the rate of complications in intramedullary nailing and its usefulness has been previously explored only in two underpowered randomized controlled trials. Thanks to the possibility to track screw placement in real-time, allowing improved screw placement, the ADAPT system could be a valid tool, in order to minimize radiation exposure, surgical time, and rate of complications.

All the patients undergoing intramedullary nailing at the Ospedale Regionale di Lugano satisfying the eligibility criteria reported at section 7.1 will be enrolled in the study and randomly allocated (allocation ratio 1:1) to receive preoperatively:

* Intramedullary nailing with ADAPT system (arm-A)
* Intramedullary nailing without ADAPT system (arm-B) Patients and physicians evaluating the results will be blinded to the assigned group.

The total number of patients enrolled will be 96 (48 arm-A, 48 arm-B). After surgery, data about duration of the procedure, intraoperative blood loss, satisfaction of the surgeon and radiation exposure time will be collected.

Fracture healing, and rate of complications (cut-through and cut out) will be evaluated during all the follow-up visits, alongside VAS and a functional evaluation of the injured hip through the Oxford Hip score.

All treatment related adverse events will be reported up to follow-up visit 4, i.e. up to 12 ± 1 months.

Every patient will be involved in the trial for 1 year. The expected time to complete the trial is 4 years: 3 years for patient enrolment and 1 year to complete the last follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary intramedullary nailing at the Ospedale Regionale di Lugano.
* Patients aged 50-85 years old.
* Patients with a BMI >18 and <35.
* Patients able to provide informed consent and follow all the study procedures as indicated by the protocol.
* Radiological evidence of proximal fracture of the femur, AO classified as 31 A1.3, 31 A2.1, 31 A2.2, 31 A2.3, 31 A3.1, 31 A3.2, 31 A3.3.

Exclusion Criteria:

* Other clinically significant concomitant disease states (e.g. renal failure, major hepatic dysfunction, life-threatening cardiovascular disease, etc..).
* Known or suspected non-compliance, drug or alcohol abuse.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
TAD (tip to apex) index at the post-operative X-Ray control prior discharge | immediately after the surgery
  The primary outcome of the study is the TAD (tip to apex) index at the post-operative X-Ray control prior discharge.
  The TAD is the tip-apex distance, which is the sum of the distance from the tip of the lag screw to the apex of the femoral head on an anteroposterior radiograph and this distance on a lateral radiograph, after controlling for magnification. The percentage of cut-outs has been correlated directly to both the severity of proximal femoral fractures and the TAD.

SECONDARY OUTCOMES:
time of the procedure | immediately after the surgery
  time
intraoperative blood loss | during the surgery
  intraoperative blood loss
intraoperative radiation time | during the surgery
  intraoperative radiation time
surgeon satisfaction on the satisfaction Numerical Rating Scale (NRS scale) | immediately after the surgery
  The satisfaction NRS is a self-assessment scale in which surgeons rate their satisfaction on an 11-point numerical scale from 0 (completely dissatisfied) to 10 (completely satisfied). The satisfaction NRS will be administered after surgery
non-union | at 6 weeks, 3 months, 6 months and 1-year
  fracture not alligned
cut-through rate | at 6 weeks, 3 months, 6 months and 1-year
  cut-through rate
cut-out rate | at 6 weeks, 3 months, 6 months and 1-year
  cut-out rate
VAS | at 6 weeks, 3 months, 6 months and 1-year
  Visual pain analogue scale, [from 0 (no pain) to 10 (worst pain)]
Oxford Hip Score, [from 0 (severe hip arthritis) to 48 ( satisfactory joint function)] | at 6 weeks, 3 months, 6 months and 1-year
  Hip function

OTHER OUTCOMES:
re-fracture rates | at 6 weeks, 3 months, 6 months and 1-year
  re-fracture rates

CONTACTS AND LOCATIONS:
Overall Officials: Christian Candrian, MD, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Christian Candrian, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No
not foreseen